CLINICAL TRIAL: NCT03165396
Title: The Appropriate Compatibility of Propofol and Sevoflurane for Orthopaedic Surgery of Patients With Mild Cognitive Impairment
Brief Title: Appropriate Compatibility of Propofol and Sevoflurane for Orthopaedic Surgery of Patients With MCI
Acronym: MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Central Clinical College of Tianjin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: szxlcyj-chen
Record Dates: First submitted 2017-05-17; First posted 2017-05-24 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2017-05

CONDITIONS: Cognitive Impairment, Mild
Keywords: mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propofol (Experimental): administrated Target Controlled Infusion （TCI）of propofol （Cp 2.0~2.5μg/ml ）for maintaining
  Interventions: Drug: Propofol
- 1.2 μg/ml Propofol (Experimental): administrated Target Controlled Infusion （TCI）of propofol （Cp 1.2 μg/ml ）combined with appropriate sevoflurane for maintaining
  Interventions: Drug: Propofol; Drug: Sevoflurane
- 0.6 μg/ml Propofol (Experimental): administrated Target Controlled Infusion （TCI）of propofol （Cp 0.6 μg/ml ）combined with appropriate sevoflurane for maintaining
  Interventions: Drug: Propofol; Drug: Sevoflurane
- Sevoflurane (Experimental): administrated 1.3 minimum alveolar concentration（MAC ） sevoflurane for maintaining
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol is the most common clinical anesthetics.
  Arms: 0.6 μg/ml Propofol; 1.2 μg/ml Propofol; Propofol
Drug: Sevoflurane — Sevoflurane is the most common clinical anesthetics.
  Arms: 0.6 μg/ml Propofol; 1.2 μg/ml Propofol; Sevoflurane

SUMMARY:
According to the inclusion and exclusion criteria, elderly patients undergoing elective orthopedic surgery were randomly divided into four groups. The different combinations of propofol and sevoflurane were used in the four groups: 1 day before surgery, after patients become wide-awake, and 3 days, 7 days, and 3 months after surgery, the patient's cognitive function was evaluated using a professional cognitive scale and other indicators. Finally, statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Elective orthopaedic surgery
* American Society of Anesthesiologists physical status: II

Exclusion Criteria:

* Neurological diseases that may affect cognitive function (e.g., subdural hematoma)
* Hypothyroidism
* Alcoholic dementia

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically cognitive function decline ：Apolipoprotein J（ApoJ） | Change from Baseline Apolipoprotein J at 7 days
  Measurement by ELISA kit

SECONDARY OUTCOMES:
Evidence of clinically cognitive function decline ：Soluble CD14（sCD14） | Change from Baseline Soluble CD14 at 7 days
  Estimating by ELISA kit
Mini mental Examination(MMSE) | preoperative 24 hours ， 7 days post surgery
  A questionnaires is used to assess the cognitive function of patients in clinical.Total range was 0~30，≦27 were considered as cognitive function decline
Montreal Cognitive Assessment（MoCA) | preoperative 24 hours ，7 days post surgery
  A questionnaires is used to assess the cognitive function of patients in clinical.Total range was 0~30，≦27 were considered as cognitive function decline.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Central Hospital of Tianjin, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes